CLINICAL TRIAL: NCT03553225
Title: Randomized, Double-blind, Placebo Controlled, Parallel Study to Evaluate the Effect of Concord Grape Extract on Vascular Function in Healthy Men and Women
Brief Title: Randomized, Double-blind, Controlled Study to Evaluate the Effect of Concord Grape Extract on Vascular Function in Healthy Men and Women
Acronym: CONCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Naturex-Dbs (Industry)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principle Investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DBS12-CRG
Record Dates: First submitted 2018-05-29; First posted 2018-06-12 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Healthy Men and Women
Keywords: vascular function; endothelial function; polyphenols; Concord Grape

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Formulation containing inert artificially colored maltodextrin, once daily, in a 2-hard capsules regimen (1g)
  Interventions: Dietary Supplement: Placebo
- Concord Grape Extract 1 (Active Comparator): 1 g Concord Grape Extract in 2 capsules
  Interventions: Dietary Supplement: Concord Grape extract 1
- Concord Grape Extract 2 (Active Comparator): 500 mg Concord Grape Extract in 2 capsules
  Interventions: Dietary Supplement: Concord Grape extract 2

INTERVENTIONS:
Dietary Supplement: Placebo — Identical formulation as the treatment consisting of colored maltodextrin using artificial colors
  Arms: Placebo
Dietary Supplement: Concord Grape extract 1 — 1 g Concord Grape extract in 2 capsules
  Arms: Concord Grape Extract 1
Dietary Supplement: Concord Grape extract 2 — 500 mg Concord Grape extract in 2 capsules
  Arms: Concord Grape Extract 2

SUMMARY:
Concord grape (Vitis Labrusca) is rich in polyphenols such as anthocyanins, flavanols, procyanidins and flavonols. Current reports investigating the effects of Concord grape (CG) consumption on cardiovascular disease (CVD) risk have provided mixed results. Studies were limited by small sample size or lacked a control arm. Moreover, subjects presented with CVD or CVD risk factors and thus to our knowledge, it remains unknown as to whether the consumption of Concord Grape (poly)phenols can maintain vascular function in healthy individuals. The aim of this study is therefore to examine both acute and chronic effects of Concord Grape on cardiovascular health by investigating whether daily consumption of Concord Grape Extract (CGE) for 12 weeks can affect biomarkers of CVD risk, including endothelial function, blood pressure and blood lipids, in young healthy men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women (pre and post-menopausal) aged 18-40 years
* Subjects are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study
* Are able to understand the nature of the study
* Able to give signed written informed consent
* Signed informed consent form

Exclusion Criteria:

* Medical history of cardiovascular disease including coronary artery disease, cerebrovascular disease and peripheral artery disease
* Hypertensive, as defined as SBP superior or equal to 140 mmHg
* Obese participants, defined as BMI superior or equal to 30 kg/m2
* Medical history of diabetes mellitus, metabolic syndrome, terminal renal failure or malignancies
* Abnormal heart rhythm (lower or higher than 60-100 bmp)
* Allergies to berries or other significant food allergy
* Subjects under medication that can affect the cardiovascular system or on vitamin/dietary supplements.
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently in a diet
* Subjects who reported participant in another study within one month before the study start
* Subjects who smoke an irregular amount of cigarettes per day
* Pregnant women or planning to become pregnant in the next 6 months
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | 12 weeks
  Determine changes in flow mediated dilation (FMD) of the brachial artery after 12 week consumption of 500 mg or 1 g of Concord grape extract vs. Placebo

SECONDARY OUTCOMES:
Changes in flow mediated dilation (FMD) of the brachial artery | 2 hours
  Determine changes in flow mediated dilation (FMD) of the brachial artery between 2 hours post consumption of 500 mg or 1 g of Concord grape extract vs. Placebo on day 0 and 2 h post consumption of 500 mg and 1 g Concard Grape extract vs. Placebo on day 84

OTHER OUTCOMES:
Changes in systolic and diastolic blood pressure (mmHg) | 12 weeks
  Determine changes in systolic and diastolic blood pressure (mmHg) at baseline and 2 hours post consumption of 500 mg and 1 g of Concord Grape extract on day 1 and day 84
Changes in heart rate (bpm) | 12 weeks
  Determine changes in heart rate (bpm) at baseline and 2 hours post consumption of 500 mg and 1 g of Concord Grape extract on day 1 and day 84
Changes in blood lipids concentration (Total, HDL and LDL, cholesterol, triglycerides) | 12 weeks
  Determine changes in blood lipids concentration (Total, HDL and LDL, cholesterol, triglycerides) after 84 days post consumption of 500 mg or 1 g Concord Grape extract vs. Placebo
Percentage (%) of participants with any treatment-related adverse events | 12 weeks
  Determine safety and tolerability of 500 mg and 1 g of Concord Grape extract vs. Placebo (%) as per any treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, Waterloo, United Kingdom

IPD SHARING:
Plan to Share IPD: No